CLINICAL TRIAL: NCT06015802
Title: Predictive Value of Serum and Tissue Molecular Markers and Imaging Features in the Invasiveness and Prognosis of Pituitary Neuroendocrine Tumors
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, director of endocrinology department, Sun Yat-sen University
Other Study IDs: 2021450
Record Dates: First submitted 2023-08-24; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Pituitary Adenoma; Neuroendocrine Tumors
MeSH Terms: conditions — Pituitary Neoplasms; Neuroendocrine Tumors | interventions — Critical Pathways

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pituitary neuroendocrine tumors: Patients with pituitary neuroendocrine tumors: pituitary adenoma was diagnosed by clinical imaging, with or without pituitary hormone secretion function was confirmed by pituitary hormone detection.
  Interventions: Other: diagnosed and treated reasonably according to the clinical guidelines and clinical pathways

INTERVENTIONS:
Other: diagnosed and treated reasonably according to the clinical guidelines and clinical pathways — The clinical data and biological specimens of the selected patients were collected, and the patients were diagnosed and treated reasonably according to the clinical guidelines and clinical pathways. The prognosis and outcome of the disease within 5 years after discharge were observed.

SUMMARY:
As the clinical manifestations of pituitary neuroendocrine tumors vary greatly, 2.7-15% of them are resistant to conventional treatments such as surgery, drug therapy and radiotherapy, and often relapse or regrow in the early postoperative period, which is invasive and has a poor prognosis. Therefore, it is important to find imaging, histological or serum molecular markers for early prediction of the invasiveness and clinical prognosis of pituitary neuroendocrine tumors. The aim of this study is to observe the changes of biomarkers and imaging features in serum or tissues of pituitary neuroendocrine tumors during the course of disease and treatment, and to explore the biomarkers and imaging features that can predict the proliferation, progression and recurrence risk of pituitary neuroendocrine tumors after medical or surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with pituitary neuroendocrine tumors: pituitary adenoma was diagnosed by clinical imaging, with or without pituitary hormone secretion function was confirmed by pituitary hormone detection.

Exclusion Criteria:

1. Previous pathological specimen suggested pituitary carcinoma.
2. always have received radiation and chemotherapy or immune and targeted therapy of the patients.
3. with known genetic syndrome can cause excessive secretion of hormones (such as Carney syndrome, McCune - Albright syndrome, multiple endocrine neoplasia type 1, acute interstitial pneumonia) patients.
4. there are ectopic neuroendocrine tumor patients.
5. within one month before the screening for major surgery, or within 3 months before screening for patients with sphenoid pituitary surgery.
6. crisis of gland function (the pituitary gland, thyroid crisis, adrenal crisis).
7. peripheral glands or other solid tumors in patients with severe disease or blood system.
8. serious organ damage such as heart, kidney, liver, etc.
9. with severe mental or nervous system disease.
10. serious high blood glucose or poorly controlled hypertension or emergency patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pituitary neuroendocrine tumors: pituitary adenoma was diagnosed by clinical imaging, with or without pituitary hormone secretion function was confirmed by pituitary hormone detection.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Disease progression or recurrence after surgery | up to 5 years
  Disease'recurrence'corresponded to tumour detection at MRI and/or hormone hypersecretion in previously cured patients, while disease'progression'indicated the increase in size of post-operative tumour remnant in nonfunctioning tumours and/or relapse of hormone hypersecretion in functioning ones

CONTACTS AND LOCATIONS:
Locations (1):
- endocrinology department of the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China